CLINICAL TRIAL: NCT07308730
Title: Randomized Controlled Trial on the Use of Pain Diary in Assessing Early Postoperative Pain Following Laparoscopic Cholecystectomy
Brief Title: Pain Diary Use After Laparoscopic Cholecystectomy
Acronym: PDP-LC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, MUHAMMED ASLAN, Graduate Student (MSc) in Surgical Nursing, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 250100; Decision No: 102 (Other: Muğla Sıtkı Koçman University Healt Sciences Ethic Committee)
Record Dates: First submitted 2025-12-17; First posted 2025-12-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cholelithiasis; Postoperative Pain
Keywords: Postoperative Pain; Daily Pain Assessment; Laparoscopic Cholecystectomy; Pain Diary
MeSH Terms: conditions — Cholelithiasis; Pain, Postoperative | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: This study uses a parallel design with two groups: an intervention group receiving the pain management protocol and a control group receiving standard care.
Masking Description: No masking is performed in this study; both participants and researchers are aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Management Intervention Group (Experimental): Participants in this group will follow the pain management protocol after laparoscopic cholecystectomy, including recording postoperative pain in a pain diary.
  Interventions: Behavioral: Postoperative Pain Management Protocol for Laparoscopic Cholecystectomy
- Control Group (No Intervention): Participants in this group will receive standard care after laparoscopic cholecystectomy. Postoperative pain will be assessed using the Visual Analog Scale (VAS) at scheduled times by nurses and researchers, and recorded accordingly

INTERVENTIONS:
Behavioral: Postoperative Pain Management Protocol for Laparoscopic Cholecystectomy — This pain management protocol is specifically tailored for patients undergoing laparoscopic cholecystectomy and combines both scheduled pharmacological analgesics and non-pharmacological pain control measures. Unlike other studies, it includes daily pain diary monitoring to objectively track patient-reported postoperative pain and recovery outcomes.
  Arms: Pain Management Intervention Group

SUMMARY:
This randomized controlled study aims to evaluate the effectiveness of using a pain diary in the assessment of early postoperative pain in patients undergoing laparoscopic cholecystectomy. Patients will be randomly assigned to a pain diary group or a control group receiving routine pain assessment. Postoperative pain intensity will be measured at predefined time points using standardized pain assessment tools. The study seeks to improve patient participation in postoperative pain evaluation without introducing additional pharmacological interventions.

DETAILED DESCRIPTION:
This is a single-center, randomized controlled trial conducted in patients undergoing elective laparoscopic cholecystectomy. Eligible patients are randomly assigned to either the intervention group or the control group using a block randomization method.

In the intervention group, postoperative pain assessment is performed using a patient-completed pain diary. The pain diary is developed based on the literature and expert opinions and is introduced to patients during the preoperative period. Patients are instructed on how to complete the pain diary, and pain intensity is recorded at rest and during movement at predefined postoperative time points.

In the control group, postoperative pain assessment is carried out using routine clinical practice with the Visual Analog Scale (VAS). Pain assessments are performed at the same postoperative time points as in the intervention group.

Additional pain-related assessments are conducted in both groups during the postoperative period. To minimize contamination between groups, patients in the intervention and control groups are followed in separate hospital rooms. Due to the visible nature of the pain diary, blinding is not feasible in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted for elective laparoscopic cholecystectomy
2. Scheduled for first-time laparoscopic cholecystectomy
3. Aged 18 years or older
4. Able to speak, read, and understand Turkish
5. Literate
6. Communicative and cooperative
7. ASA score of 1, 2, or 3
8. Expected to stay at least 24 hours in the hospital post-surgery
9. Capable of understanding study instructions
10. Willing to participate voluntarily

Exclusion Criteria:

1. Prolonged stay in the recovery unit due to extended effects of general anesthesia
2. Admission to intensive care unit postoperatively
3. Having chronic pain and receiving treatment for it
4. Being a cancer patient
5. Having a writing disability
6. Inability to communicate
7. Having cognitive, affective, verbal, visual, or auditory impairments
8. Diagnosed psychiatric disorders such as anxiety or depression and using related medications
9. Choosing to withdraw from the study after giving consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity and Pain Diary vs. VAS Comparison | During the first 48 hours post-surgery (measurements at 2, 4, 6, 12, 16, 20, 24, 32, and 48 hours postoperatively)
  The primary outcome measure involves postoperative pain intensity recorded by patients in the intervention group using a daily pain diary, compared to routine clinical VAS measurements in the control group. Measurements will be taken at 2, 4, 6, 12, 16, 20, 24, 32, and 48 hours post-surgery. Additionally, short pain inventories at 24 and 48 hours and VAS-based satisfaction evaluation before discharge will be performed.

SECONDARY OUTCOMES:
Postoperative Pain Intensity | During the first 48 hours post-surgery (measurements at 2, 4, 6, 12, 16, 20, 24, 32, and 48 hours postoperatively)
  Postoperative pain intensity will be assessed using a 0-10 Likert scale (VAS). In the intervention group, patients will record their pain in a daily pain diary at scheduled times, while in the control group, routine clinical VAS measurements will be performed. Additionally, short pain inventories at 24 and 48 hours and VAS-based satisfaction evaluation before discharge will be conducted

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah K KÖSE, Study Director — Muğla Sıtkı Koçman University / Faculty of Health Sciences Department of Nursing
Locations (1):
- Menteşe State Hospital, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The specific individual patient data collected in this study include patient first and last names, signed informed consent forms, socio-demographic information (age, gender, etc.), medical history, and postoperative pain diary data. These data will be used solely for research purposes and shared in accordance with confidentiality principles
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual patient data and supporting information will be accessible from the date patients provide informed consent prior to surgery, throughout the data collection period, and for at least 5 years following study completion, stored in accordance with confidentiality principles
Access Criteria: Individual patient data and supporting information will be accessible only to the study research team. The research team will have access to patient names, surnames, socio-demographic information, medical history, and pain diary data via a secure, password-protected electronic database. The data will be used solely for study purposes and will not be shared with third parties